CLINICAL TRIAL: NCT04444193
Title: Safety and Efficacy Study of Durvalumab in Combination With Lenvatinib in Participants With Advanced and Recurrent Endometrial Carcinoma--DULECT Trial
Brief Title: Durvalumab and Lenvatinib in Participants With Advanced and Recurrent Endometrial Carcinoma
Acronym: Dulect2020-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHFMIH-IIT-2020-0005
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — durvalumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab and Lenvatinib (Experimental): Combination therapy of Lenvatinib 80-120mg daily orally and durvalumab 1500mg by IV infusion every 4 weeks
  Interventions: Drug: Durvalumab; Drug: Lenvatinib Oral Product

INTERVENTIONS:
Drug: Durvalumab — Anti-PD-L1 Monoclonal Antibody
  Other Names: Durvalumab injection
Drug: Lenvatinib Oral Product — Lenvatinib (Lenvima, Eisai China) is a novel angiogenesis inhibitor which targets vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT
  Other Names: LENVIMA

SUMMARY:
This study will evaluate the safety and efficacy of durvalumab in combination with lenvatinib in participants with advanced and recurrent endometrial carcinoma.The primary hypothesis of this study are that patients with advanced and recurrent endometrial carcinoma could benefit from durvalumab plus lenvatinib with respect to: 1)Progression Free Survival (PFS) ; 2) Objective Response Rate (ORR); and Overall survival (OS). The investigators design a clinical study to explore whether the combination above as a treatment in patients with advanced and recurrent endometrial carcinoma could prolong PFS and to analyze potential immune biomarker of therapeutic response.

DETAILED DESCRIPTION:
The combination of Lenvatinib and Programmed death-ligand 1 (PD-L1) blocking has great potential in the treatment of advanced and recurrent endometrial cancer. This trial is designed as a prospective, open label study for 20 patients with advanced (recurrent, refractory or metastatic) endometrial cancer, including carcinosarcoma of the uterus. The aim is to investigate the efficacy of the combination therapy of Lenvatinib 80-120mg daily orally and durvalumab 1500mg by IV infusion every 4 weeks in terms of progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of screening and female.
* Histologically confirmed diagnosis of epithelial endometrial carcinoma.
* Patient must have endometrial cancer in one of the following categories:

  * Newly diagnosed Stage III disease (measurable disease per RECIST 1.1 following surgery or diagnostic biopsy),
  * Newly diagnosed Stage IV disease (with or without disease following surgery or diagnostic biopsy)
  * Recurrence of disease where the potential for cure by surgery alone or in combination is poor.
* Not eligible for hormonal therapy (because of negative hormone receptor/poor differentiation, or after failure of hormonal therapy).
* Naïve to first line systemic anti-cancer treatment. For patients with recurrent disease only, prior chemotherapy is allowed only if it was administered in the adjuvant setting and there is at least 12 months from date of last dose of chemotherapy administered to date of subsequent relapse
* Adequate organ system function as measured within 28 days prior to administration of study treatment, as defined below:

Haemoglobin ≥ 10.0 g/dL, with no blood transfusion in the past 28 days. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L Platelet count ≥ 100 x 10^9/L Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (not applicable to Gilbert's syndrome) Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x ULN unless liver metastases are present in which case they must be ≤ 5x ULN Patients must have creatinine clearance estimated of ≥51 mL/min estimated using the Cockcroft-Gault equation or 24 hr urine clearance.

Exclusion Criteria:

* Any previous treatment with a PD1 or PD-L1 inhibitor
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* History of leptomeningeal carcinomatosis, symptomatic uncontrolled brain metastases (≤2mg/ day corticosteroids started ≥4 weeks prior to treatment is accepted) and spinal cord compression (unless received definitive treatment and clinically stable for 28 days) .
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active tuberculosis (TB; Bacillus tuberculosis).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to Cycle 1, Day 1.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1, Day 1.
* Has severe hypersensitivity (≥Grade 3) to Durvalumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3 years
  Defined as time from randomisation to first progression by investigator assessment using modified RECIST 1.1 or death (by any cause in the absence of progression)
Objective Response Rate (ORR) | Up to 3 years
  Objective response rate is defined as the proportion of patients with measurable disease at baseline who have confirmed complete response (CR) or partial response (PR) as determined by the Investigator at local site

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  Defined as the time from randomisation to death due to any cause
Percentage of Participants who Experience an Adverse Event (AE) | Up to 1 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Wan, MD.,Ph.D, Study Chair — Shanghai First Maternity and Infant Hospital; Huan Tong, Principal Investigator — Shanghai First Maternity and Infant Hospital